CLINICAL TRIAL: NCT05470439
Title: Pharmacist-CHW Team to Improve Medication Adherence and Reduce Hypertension
Brief Title: My Interprofessional Care Team for Adherence and Research Engagement Disparities
Acronym: MI-CARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: University of Massachusetts, Amherst (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: R01HL151772 (NIH)
Record Dates: First submitted 2022-07-14; First posted 2022-07-22 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Medication Adherence; Hypertension
Keywords: Pharmacist, CHW, Hypertension, Adherence, FQHC
MeSH Terms: conditions — Medication Adherence; Hypertension

STUDY DESIGN:
Intervention Model Description: MI-CARE is an innovative, tailored coordinated care intervention by pharmacist-community health worker (CHW) team derived from a previous research and a clinical pilot implementation. MI-CARE will identify and address individual, clinical, social-cultural and structural barriers to medication adherence and hypertension management. MI-CARE consists of an initial individualized needs assessment (Baseline). During Month 1 and Month 2, pharmacist-CHW team will deliver a tailored intervention including an individualized medication chart, preferred adherence aids, hypertension therapy optimization, tailored education based on medication beliefs, tools to combat social stressors, and referrals for structural barriers such as food insecurity, transportation, and drug costs. Tailored family/care partner participation and telehealth visits will be provided when needed during this time. A booster visit to assess patient progress and reinforce intervention components will occur at Month 2.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MI-CARE Intervention (Experimental): Pharmacist-community health worker team providing coordinated care tailored to high-risk patients with hypertension. MI-CARE intervention participants will meet with the pharmacist-CHW team for medication optimization and tailored case management. Pill counts will be completed to assess adherence and BP will be measured at each visit to guide antihypertensive medication optimization and provide feedback to participants about their adherence and BP control. Intervention visits will be followed by a booster one month later.
  Interventions: Behavioral: My Interprofessional Care team for Adherence and Research Engagement (MI-CARE)
- Waitlist Control (No Intervention): Participants enrolled in this arm will receive usual medical care

INTERVENTIONS:
Behavioral: My Interprofessional Care team for Adherence and Research Engagement (MI-CARE) — MI-CARE is an innovative, tailored coordinated care intervention by pharmacist-community health worker (CHW) team derived from a previous research and a clinical pilot implementation. MI-CARE will identify and address individual, clinical, social-cultural and structural barriers to medication adherence and hypertension management. MI-CARE consists of an initial individualized needs assessment (Baseline). During Months 1-2, pharmacist-CHW team will deliver a tailored intervention including an individualized medication chart, preferred adherence aids, hypertension therapy optimization, tailored education based on medication beliefs, tools to combat social stressors, and referrals for structural barriers such as food insecurity, transportation and drug costs. Tailored family/care partner participation and telehealth visits will be provided when needed during this time. A booster visit to assess patient progress and reinforce intervention components will occur at Month 2.
  Arms: MI-CARE Intervention

SUMMARY:
MI-CARE is an innovative coordinated care team intervention to improve medication adherence and blood pressure derived from research findings that build on existing clinical practice. Designed with an eye toward sustainability, MI-CARE incorporates billable pharmacist and CHW services for patients with low medication adherence and high burdens of chronic illness and preventable consequences. MI-CARE offers interprofessional team care with comprehensive expertise and complementary skill sets that mitigate the silo effect of specialized medicine to deliver primary care to diverse, high-risk populations experiencing disparities in hypertension.

DETAILED DESCRIPTION:
MI-CARE is a practice-based randomized controlled trial (RCT) to test the effectiveness of a comprehensive, individually- and culturally-tailored intervention for high-risk patients with hypertension, polypharmacy, and low adherence. MI-CARE leverages the specialized expertise of a clinical pharmacist together with a community health worker (CHW) who will serve as a cultural broker and patient navigator to address individual, clinical, social-cultural, and structural barriers to adherence.

This comprehensive and tailored, coordinated care intervention aims to improve medication adherence and hypertension outcomes among African-American, Latino, and Vietnamese immigrant patients. The proposed practice-based RCT is designed to meet the following specific aims:

Aim 1: Implement MI-CARE, an innovative, tailored adherence intervention delivered by a pharmacist and CHW team.

Aim 2: Determine the short- and long-term effectiveness of MI-CARE by assessing pre- to post-intervention changes in a) medication adherence (proximal outcome) and blood pressure (BP, distal outcome), and b) other comorbid health outcomes (e.g., HbA1c, BMI) using a randomized controlled trial.

Aim 3: Identify factors associated with MI-CARE effectiveness including a) tailored intervention features, b)medication beliefs, c) barriers to adherence, d) intervention dose, e) health literacy and f) cultural group.

The investigators will follow an intention-to-treat randomized design using a waitlist control with 230 African-American, and Latino patients with hypertension and low (<85%) medication adherence. Data collection via pill count, self-report, electronic health record, and clinical measures will assess medication adherence, BP, and other factors at baseline (pre-intervention) and at 6 months post-intervention.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 18 years;
2. self-report cultural identity as African-American, or Latino;
3. speak English, or Spanish;
4. have medication-treated hypertension;
5. use ≥5 chronic medications;
6. have hypertension medication adherence <85%; and
7. able to provide informed consent.

Exclusion Criteria:

1. if project staff conclude that a candidate participant is unable to comprehend the informed consent process (because he/she offers an inappropriate response to consent questions); or
2. if the candidate is hostile or unwilling to follow project protocols.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Objectively measured medication adherence (pill count) | Month 6
  The investigators will use dosage information from the pill bottle and refill history to calculate percentage adherence (the number of pills taken / the number of pills that should have been taken x 100). All chronic oral medications in current use will be counted. Percent adherence rates for each medication will be calculated as well as the mean adherence averaged across all chronic oral medications.
Self-reported medication adherence (survey) | Month 6
  Medication Adherence Report Scale-5 (MARS-5) with 5-point Likert scale will be used (Minimum Value: 1; Maximum Value 5); Range of score (cumulative): 5(worst) - 25(best)
Blood Pressure | Month 6
  Systolic and diastolic blood pressure measured by a calibrated, automated sphygmomanometer

SECONDARY OUTCOMES:
HgbA1c | Month 6
  Hemoglobin A1c for participants with concurrent diabetes will be collected from electronic health record
Weight | Month 6
  Participant's weight will be collected from electronic health record
Body Mass Index (BMI) | Month 6
  BMI calculated using participant's height and weight will be collected from electronic health record
Lipid | Month 6
  Lipid panel including low-density lipoprotein (LDL) cholesterol level will be collected from electronic health record
Statin use | Month 6
  Use of statin medication for participants with dyslipidemia or clinical atherosclerotic cardiovascular disease (or risk >7.5%) will be collected from electronic health record

CONTACTS AND LOCATIONS:
Overall Officials: Jeannie K Lee, PharmD, Principal Investigator — University of Arizona College of Pharmacy
Locations (1):
- Caring Health Center, Inc., Springfield, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No